CLINICAL TRIAL: NCT04376216
Title: Prednisolon Behandling Ved Akut Interstitiel Nefritis - et Randomiseret, Prospektivt Studie
Brief Title: Prednisolone Treatment in Acute Interstitial Nephritis
Acronym: PRAISE
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Region MidtJylland Denmark (Other)
Collaborators: Aarhus University Hospital (Other); Odense University Hospital (Other)
Responsible Party: Principal Investigator, Frank Mose, Associate professor, Region MidtJylland Denmark
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FHM-1-2017
Record Dates: First submitted 2020-04-27; First posted 2020-05-06 (Actual); Last update posted 2020-12-30 (Actual); Status verified 2020-12

CONDITIONS: Acute Tubulo-Interstitial Nephritis
Keywords: Acute Tubulo-Interstitial Nephritis; Prednisone
MeSH Terms: conditions — Acute Tubulointerstitial Nephritis | interventions — Prednisone; Prednisolone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control (No Intervention): No treatment
- Prednisone (Active Comparator): Oral prednisone. Starting dose of 60 mg with tapering for 2 months
  Interventions: Drug: Prednisone

INTERVENTIONS:
Drug: Prednisone — 60 mg with dose tapering over 2 months
  Other Names: Prednisolone
  Arms: Prednisone

SUMMARY:
A Prospective randomized trial with a primary objective to investigate the effect ofprdenisolone treatment in acute interstitial nephritis

ELIGIBILITY:
Inclusion Criteria:

* Biopsy verified AIN
* Clinical suspicion of AIN
* Age > 18 years
* One of following criteria:

  * Plasma creatinine > 120 µmol/L or
  * Plasma creatinine increase > 30 µmol/L or increase > 50 % of baseline plasma creatinine
* Fertile women are included

Exclusion Criteria:

* No ability to give informed consent
* Immunosuppressive treatment (including prednisolone) within 3 months before biopsy
* Autoimmune disease
* Prednisolone intolerance
* Pregnancy or lactation
* Active cancer (except basal cell carcinoma)
* Short life expectancy (< 6 months)
* CKD stage IV-V
* AIN secondary to or accompanied by glomerulonephritis, sarcoidosis or inherited interstitial renal disease
* Previous participation Withdrawal criteria
* Development of exclusion criterion
* Withdrawal of consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2017-09-01 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2027-09-01 (Estimated)

PRIMARY OUTCOMES:
eGFR | 3 months
  Kidney function

SECONDARY OUTCOMES:
eGFR | 12 months
  Kidney function
Urinary biomarkers | at inclusion and after3 and 12 months
  NGAL, NAG, KIM-1, TIMP-2, IGFBP7, IL-6, IL-18 and MCP-1 are the biomarkers that the investigators plan to analyze
Pathology | At inclusion
  Re-evaluation of renal biospies performed at time of inclusion. This evaluation includes the use of routine and special staining for inflammation, fibrosis and tubular damage. The analysis includes an estimation of predictive value of histological scoring on treatment response and prognosis
Need for renal replacement therapy | 3 and 12 months
  Dialysis need
Plasma glucose or hemoglobin A1C | 3 and 12 months
  Development of diabetes (safety)
Treatment delay | At inclusion
  In the prednisolone group the importance of "treatment delay" is analyzed. Treatment delay is defined as follows:
  * Days form first symptoms to inclusion in this project
  * Days from first contact to the Danish health care system to inclusion in this project
  * Days from first contact to a nephrology department to inclusion in this project
Infections (number of events) | 3 and 12 months
  Safety
Admissions (number of events) | 3 and 12 months
  Safety

CONTACTS AND LOCATIONS:
Overall Officials: Jesper N Bech, MD, Study Chair — Region MidtJylland Denmark
Locations (1):
- Godstrup Hospital, Herning, Denmark

IPD SHARING:
Plan to Share IPD: Undecided
Will be decided

REFERENCES:
- [Derived] Mose FH, Birn H, Hoffmann-Petersen N, Bech JN. Prednisolone treatment in acute interstitial nephritis (PRAISE) - protocol for the randomized controlled trial. BMC Nephrol. 2021 May 1;22(1):161. doi: 10.1186/s12882-021-02372-4. PMID 33933012